CLINICAL TRIAL: NCT04691960
Title: A Pilot Study of Ketogenic Diet and Metformin in Glioblastoma: Feasibility and Metabolic Imaging
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1604017166
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Diet, Ketogenic; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Ketogenic Diet (Experimental)
  Interventions: Other: Ketogenic Diet; Drug: Metformin

INTERVENTIONS:
Other: Ketogenic Diet — Ketogenic diet is high-fat, low carbohydrate diet. Ketogenic diet will be maintained on a continuous basis. The diet will begin at an approximately 3:1 fat to carbohydrate + protein ratio for 5 days. If the patient does not show urine ketosis (1.5 mmol/L or 27.0 mg/dL), the ketosis diet will be advanced to approximately 4:1 ratio for 5 days. If the patient still does not attain ketosis a 24 hour fast will be done to promote ketosis. The diet will encourage at least 30 ml per day of Medium Chain Triglycerides (MCT) oil to enhance ketosis.
Drug: Metformin — Metformin will be administered as a single 850 mg dose P.O. at Week 8, then titrated up to 850 mg P.O. BID at Week 10, and then 850 mg T.I.D. at Week 12, as tolerated.

SUMMARY:
This clinical trial is for men and women with high-grade gliomas. Glucose (sugar) is thought to be a contributor to tumor growth. The ketogenic diet (a high fat, low carbohydrate diet) and metformin (a drug approved by the Food and Drug Administration to treat type 2 diabetes) are both known to lower blood glucose levels. The purpose of the study is to evaluate the tolerability of a ketogenic diet in conjunction with metformin and whether maintaining and the diet with metformin will have any effect on participants. Participants will prepare their own meals with the help of a nutritionist. Participants will continue on treatment as long as they are responding to therapy and not experiencing unacceptable side effects

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed high-grade glioma (e.g. glioblastoma, gliosarcoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed glioma or other anaplastic gliomas).
2. Patients must have an MRI performed within 21 days prior to beginning the study diet and on a fixed dose of steroids for at least 5 days. If the steroid dose is increased between the date of imaging and registration, a new baseline MR/CT is required.
3. Patients must not have been exposed to bevacizumab.
4. Patients cannot be taking insulin or other oral hypoglycemic. Must be at least 6 weeks from last oral hypoglycemic or insulin.
5. Must not have known type 1 or type 2 diabetes and expected to need either insulin and/or an oral hypoglycemic agents within the next 6 months.
6. Patients must be >18 years old.
7. Karnofsky performance status >60%.
8. Life expectancy of greater than 12 weeks.
9. Patients must have normal organ and marrow function as defined below:

   * Leukocytes >3,000/mcL
   * Absolute neutrophil count >1,000/mcL
   * Platelets >100,000/mcL
   * Total bilirubin <2.0 X institutional upper limit of normal (unless known to have Gilbert's Disease)
   * AST (SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
   * Serum Glucose: < 200 mg/dL
   * Creatinine < 1.5 mg/dL (for males), < 1.4 mg/dL (for females), or within normal lab limits OR
   * Creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
10. Patients must not have any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy
11. Patients having undergone recent resection or progressive tumor will be eligible as long as all of the following conditions apply:

    1. They have recovered from the effects of surgery.
    2. On a steroid dosage that has been stable for at least 5 days.
    3. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease postoperatively, a MRI should be done:

       * No later than 96 hours in the immediate post-operative period or
       * At least 4 weeks post-operatively, and
       * Within 14 days of registration, and
       * If the 96-hour scan is more than 21 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI is required on a stable steroid dosage for at least 5 days.
12. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who are receiving any other investigational agents.
2. Patients who have had prior therapy with bevacizumab and/or other VEGF inhibitors.
3. Patients who are taking insulin or other oral hypoglycemic. Must be at least 6 weeks from last oral hypoglycemic or insulin.
4. History of allergic reactions attributed to metformin.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, diabetes requiring oral hypoglycemic drugs and/or insulin, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients known to have a malignancy that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except nonmelanoma skin cancer or carcinoma in-situ in the cervix).
7. The effects of a Ketogenic diet or metformin on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
8. Patients with current alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Ability to achieve and maintain ketosis | Through study completion (an average of 8 months)
  Proportion of patients who can obtain and maintain a ketogenic state (of 1.5 mmol/L or 27.0 mg/dL)
Tolerability of metformin | Through study completion (an average of 8 months)
  Proportion of patients who can tolerate Metformin in the setting of the ketogenic diet (as assessed by standard CTC criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fine, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided